CLINICAL TRIAL: NCT04598555
Title: A Multi-centre Multi-country Prospective obseRvatIonal Study on Patterns of Care of Mild Asthmatic patiEnts
Brief Title: Study on Patterns of Care in Mild Asthmatic Patients
Acronym: PRIME
Status: Completed | Type: Observational
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLI-01535AA0-01
Record Dates: First submitted 2020-10-12; First posted 2020-10-22 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The PRIME study is an observational, Real World Evidence study designed to collect the type of treatments that are currently prescribed to patients with mild asthma and to collect relevant clinical data that could reflect the control of the disease over a 6-month observational period according to the standard clinical practice.

DETAILED DESCRIPTION:
Outpatients attending the hospital clinics/study centres will be recruited. Patients with mild asthma treated by Step 1 or step 2 treatments according to GINA report will be recruited. A total of approximately 1200 patients will be enrolled. Patients will be followed-up during a 6-month observational period according to standard practices.

ELIGIBILITY:
Inclusion Criteria:

* Adult subject (aged ≥ 18 years) up to 75 years
* Subject with confirmed asthma diagnosis
* Subject in treatment for mild asthma with Step 1 or Step 2 according to GINA report
* Subject with written privacy and study informed consent

Exclusion Criteria:

* Subject enrolled in experimental (interventional) clinical trials, or receiving experimental treatments in the prior 3 months
* Known pregnant or breast-feeding subject
* Subject unable to understand and autonomously fill in questionnaires
* Subject unable to use electronic devices to fill in e-diary, or without compatible electronic devices with access to the Internet
* Subject who had asthma exacerbation(s) in the past 4 weeks prior to study entry
* Subject with confirmed Chronic Obstructive Pulmonary Disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mild asthma patients treated by step 1 or 2 treatments according to GINA report
Sampling Method: Non-Probability Sample
Enrollment: 981 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
To describe the real-world patterns of treatment of subjects with mild asthma during a 6-month observational period. | 6-months period
  Frequency of asthma treatments for asthma management, regardless the duration:
  * by active substance
  * by drug class
  * distinguishing between "controller" and "reliever" treatments
To describe the real-world patterns of treatment of subjects with mild asthma during a 6-month observational period. | 6-months period
  Frequency of subjects experiencing asthma treatment switches, step-ups and step-downs during the observation period, along with the description of pattern of switch (in terms of sequence of treatments over time)
To describe the real-world patterns of treatment of subjects with mild asthma during a 6-month observational period. | 6-months period
  Frequency of treatment posology, stratified by type of asthma treatment
To describe the real-world patterns of treatment of subjects with mild asthma during a 6-month observational period. | 6-months period
  Duration of asthma treatments (in months):
  * overall
  * by drug class (i.e., any switch to drugs within the same class will be considered as a continuation of the treatment) and by active substance (i.e., any dose adaptation will be considered as a continuation of the same drug). This will be adapted according to data availability.

SECONDARY OUTCOMES:
To describe the Socio-demographics data of subjects with mild asthma at enrolment visit | At enrolment
  BMI in kg/m^2
To describe the clinical characteristics of subjects with mild asthma at enrolment visit | At enrolment
  Lifestyle and smoking habits data description
To describe the Daytime and night-time symptoms of subjects with mild asthma at enrolment visit | At enrolment
  Frequency of daytime and night-time symptoms
To describe the Daytime and night-time symptoms of subjects with mild asthma at enrolment visit | At enrolment
  Type of daytime and night-time symptoms
To describe the Asthma Diagnosis of subjects with mild asthma at enrolment visit | At enrolment
  Time from first Asthma Diagnosis
To describe the Asthma Diagnosis of subjects with mild asthma at enrolment visit | At enrolment
  Type of diagnosis strategy
To describe the asthma exacerbations of subjects with mild asthma at enrolment visit | At enrolment
  Asthma exacerbations history data description
To describe the prior asthma treatment of subjects with mild asthma at enrolment visit | At enrolment
  Type of prior Asthma treatments description
To describe the clinical characteristics of subjects with mild asthma at enrolment visit | At enrolment
  Skin Prick test data description
To describe the evolution of lung function parameters (FEV1 (L)) during the 6-month observational period | At enrolment and at 6-month
  Spirometry results at enrolment and at 6-month follow-up visit (according to sites' standard practice): measurement of Forced Expiratory Volume in 1 second (FEV1) in L
To describe the evolution of lung function parameters (FEV1 (%)) during the 6-month observational period | At enrolment and at 6-month
  Spirometry results at enrolment and at 6-month follow-up visit (according to sites' standard practice): measurement of FEV1 predicted value in %,
To describe the evolution of lung function parameters (FVC (L)) during the 6-month observational period | At enrolment and at 6-month
  Spirometry results at enrolment and at 6-month follow-up visit (according to sites' standard practice): Forced Vital Capacity (FVC) in L
To describe the evolution of lung function parameters (FVC (%))during the 6-month observational period | At enrolment and at 6-month
  Spirometry results at enrolment and at 6-month follow-up visit (according to sites' standard practice): measurement of FVC % predicted
To describe the evolution of lung function parameters (FEV1/FVC ratio) during the 6-month observational period | At enrolment and at 6-month
  Spirometry results at enrolment and at 6-month follow-up visit (according to sites' standard practice): measurement of FEV1/FVC ratio in %
To describe subjects' level of asthma symptoms control by means of the Asthma Control Test (ACT) during the 6-month observational period | At enrolment and at 6-month
  ACT score. ACT is a 5-point scale (for symptoms and activities: 1=all the time to 5= not at all; for asthma control rating: 1=not controlled at all to 5=completely controlled). ACT scores range from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control. An ACT score >19 indicates well-controlled asthma.
To describe subjects' level of asthma symptoms control by means of the Asthma Control Questionnaire (ACQ-5) during the 6-month observational period | At enrolment and at 6-month
  ACQ-5 score. ACQ-5 is a 7-point scale (0=no impairment, 6= maximum impairment) and scores range between 0 (totally controlled) and 6 (severely uncontrolled).
To describe the occurrence of asthma exacerbations during the 6-month observational period | 6-months period
  Number of Asthma exacerbations during the 6-month observational period (seriousness, severity, relatedness to the treatment product, start date and end date (duration will be calculated during data analysis), outcome, action taken with respect to drug and other treatments used to treat exacerbations)
To describe the utilization of healthcare resources in subjects with mild asthma during the 6- month observational period | 6-months period
  Number of Inward/Day-hospital hospitalizations, emergency room accesses and GP/outpatient specialist visits
To describe the utilization of healthcare resources in subjects with mild asthma during the 6- month observational period | 6-months period
  Number and type of tests and exams per subject
To describe the utilization of healthcare resources in subjects with mild asthma during the 6- month observational period | 6-months period
  Duration of Inward/Day-hospital hospitalizations
To describe the subjects' quality of life by means of the Mini Asthma Quality of Life Questionnaire (MiniAQLQ) during the 6-month observational period | At enrolment and at 6-month
  MiniAQLQ scores. The MiniAQLQ is a 7-point Likert scale (7 = not impaired at all - 1 = severely impaired) and scores range 1-7, with higher scores indicating better quality of life.
To describe the occurrence of adverse drug reactions (ADRs) in subjects with mild asthma during the 6-month observational period. | 6-month
  Only Adverse Drug Reactions (ADRs) to any asthma medication occurred during the 6-month observational period will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Eva Topole, Dr, Study Director — CHIESI Clinical Program Leader
Locations (59):
- Germany (11):
  - DE-008 Lungenarztpraxis Hellersdorf, Berlin
  - DE-003 Praxis Pneumologie und Allergologie Dr. Ginko, Bonn
  - DE-005 Praxis für Pneumologie und Innere Medizin, Fürstenwalde
  - DE-006 Studieninstitut des Pneumologicums Halle, Halle
  - DE-001 Salvus - Klinische Studien GmbH, Leipzig
  - DE-007 POIS Leipzig GbR, Leipzig
  - DE-004 Fortbildungs- und Studienzentrum Innere Medizin Marburg GbR, Marburg
  - DE-009 Praxis Dr. Jansen, Menden
  - DE-012 Pneumologisch-Internistische Gemeinschaftspraxis Elisenhof, Munich
  - DE-010 Studienzentrum Dr. Schlenska, Peine
  - DE-002 RespiRatio / Lungenpraxis Schleswig, Schleswig
- Italy (23):
  - IT-028 Fisiopatologia Respiratoria Ospedale Ecclesiastico Miulli, Acquaviva delle Fonti
  - IT-026 SOSD Allergologia A.O.U. Ospedali Riuniti, Ancona
  - IT-005 UO Allergologia Ospedale S.Maria della Speranza, Battipaglia
  - IT-019 UOC Pneumologia Ospedale Bellaria, Bologna
  - IT-008 Pneumologia Policlinico Universitario Mater Domini, Catanzaro
  - IT-006 SC MAR Univ A.O.U. Ospedali Riuniti Foggia, Foggia
  - IT-001 UOC Pneumologia Fondazione Cà Granda Ospedale Maggiore Policlinico, Milan
  - IT-007 Malattie Apparato Respiratorio A.O.U. Modena Policlinico, Modena
  - IT-025 Allergologia e Immunologia clinica Policlinico Casula A.O.U. Cagliari, Monserrato
  - IT-012 UOC Clinica Pneumologica A.O. dei Colli P.O. Monaldi, Napoli
  - IT-016 SSD Intertiziopatie e Malattie del Polmone A.O.U. San Luigi Gonzaga, Orbassano
  - IT-010 Medicina del Lavoro, Mal.Respiratorie e Tossicologia Azienda Ospedaliera, Perugia
  - IT-013 UO Pneumologia A.O.U. Pisana P.O. Cisanello, Pisa
  - IT-015 UOC Pneumologia Policlinico Univ. A. Gemelli, Roma
  - IT-020 UOC Pneumologia A.O.U. Sant'Andrea, Roma
  - IT-009 Pneumologia Clinica e Interventistica AOU Policlinico Universitario stabilim San Pietro, Sassari
  - IT-021 Servizio Pneumologia PTA Ospedale Busacca, Scicli
  - IT-024 Allergologia Casa della Salute, Scilla
  - IT-029 Malattie Respiratorie e Trapianto Polmonare A.O.U. Senese Policlinico Le Scotte, Siena
  - IT-017 Pneumologia Riabilitativa ICS Maugeri, Telese Terme
  - IT-022 Pneumologia Univ. A.O.U. Città della Salute e della Scienza, Torino
  - IT-003 UO Pneumologia Riabilitativa ICS Maugeri, Tradate
  - IT-018 USD Allergologia AOUI Policlinico Rossi, Verona
- Poland (15):
  - PL-012 Centrum Medyczne Pratia, Bydgoszcz
  - PL-018 Prywatny Gabinet Ewa Gawrońska-Ukleja, Bydgoszcz
  - PL-010 M2M Badania Kliniczne, Chorzów
  - PL-015 Prywatny gabinet Pulmonologiczny at premises of Amicmed Medical Center, Grudziądz
  - PL-005 Centrum Medyczne ALL-MED, Krakow
  - PL-001 Poradnia Alergologii i Chorób Płuc, SPZOZ Uniwersytecki Szpital Kliniczny nr 1 im Norberta Barlickiego, Lodz
  - PL-013 SNZOZ Poradnia Specjalistyczna MedMed, Ul. Brzechwy 7a, Lodz
  - PL-017 Gabinet Pulmonologiczny, Lodz
  - PL-004 CDT Medicus, Lubin
  - PL-009 Centrum Alergologii Sp. z o. o, Lublin
  - Pl-006 Ppl Ps Magmed, Radom
  - PL-014 Indywidualna Specjalistyczna Praktyka Lekarska Marzenna Tarnowska-Matusiak, Szczecin
  - PL-016 NZOZ Poradnia Chorób Płuc i Alergologii, Słupsk
  - PL-003 Praktyka lekarska Marzena Justyna Mierzejewska, Warsaw
  - PL-011 Lekarze Specjaliści J.Małolepszy i Partnerzy, Wroclaw
- Spain (10):
  - ES-005, Badalona
  - ES-009 Hospital de la Santa Creu i Sant Pau, Barcelona
  - ES-014 Hospital El Pilar, Barcelona
  - ES-002 Hospital Universitario La Princesa, Madrid
  - ES-004 'Hospital Universitario La Paz, Madrid
  - ES-008 Fundación Jiménez Díaz, Madrid
  - ES-010 Hospital Costa del Sol, Málaga
  - ES-007 Complejo asistencial Universitario de Salamanca, Salamanca
  - ES-11 Hospital Universitario Marqués de Valdecilla, Santander
  - ES-003 Hospital Universitario Dr. Peset, Valencia

IPD SHARING:
Plan to Share IPD: No